CLINICAL TRIAL: NCT03242863
Title: Strategies to Moderate Energy Intake for the Prevention of Obesity in Children
Brief Title: Effect of Varying Proportions of Low and High Energy Dense Foods Over 5 Days in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ChildFood503; R01DK082580 (NIH)
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): Baseline proportions of high and low energy dense foods.
  Interventions: Other: Food proportionality
- Addition (Experimental): Increased portion of low energy dense foods.
  Interventions: Other: Food proportionality
- Substitution (Experimental): Increased portion of low energy dense foods substituted for equal portion of foods higher in energy density.
  Interventions: Other: Food proportionality

INTERVENTIONS:
Other: Food proportionality — Proportions of high and low energy dense foods manipulated

SUMMARY:
In this study, the investigators will vary the proportions of high- and low-energy-dense foods served to preschool children at all meals and snacks during three 5-day periods. In the three experimental conditions, the same foods will be served; only the amounts and proportions of foods will be varied. In the Baseline condition, typical proportions of age-appropriate foods will be served. In the Addition condition, the portion sizes of low-energy-dense foods will be increased, and in the Substitution condition, the portions of low-energy-dense foods will be increased by replacing an equivalent amount of foods higher in energy density. The primary aim is to determine the effect on children's energy intake of varying the proportion of low- and high-energy-dense foods served, either by addition or substitution, over 5 days. It is hypothesized that children will consume less energy when they are served meals in which low-energy-dense foods are substituted for foods higher in energy density over 5 days and that children will consume more energy when served meals to which low-energy-dense foods are added. Additionally, we will test the hypothesis that daily energy intake in the three conditions will begin to converge across the 5-day period.

ELIGIBILITY:
Inclusion Criteria:

* Attending one of the designated daycare centers

Exclusion Criteria:

* Food Allergies
* Food restrictions
* Health Issues that Preclude Participation
* Not available for duration of the study

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Rolls, PhD, Principal Investigator — Penn State University
Locations (1):
- Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Rolls BJ, Roe LS, Keller KL. Children's Energy Intake Generally Increases in Response to the Energy Density of Meals but Varies with the Amounts and Types of Foods Served. Am J Clin Nutr. 2024 Jan;119(1):185-195. doi: 10.1016/j.ajcnut.2023.10.019. Epub 2023 Oct 27. PMID 37890673
- [Derived] Roe LS, Keller KL, Rolls BJ. Food Properties and Individual Characteristics Influence Children's Intake Across Multiple Days of Weighed Assessments in Childcare Programs. J Nutr. 2023 May;153(5):1646-1655. doi: 10.1016/j.tjnut.2023.03.025. Epub 2023 Mar 24. PMID 36965692
- [Derived] Roe LS, Sanchez CE, Smethers AD, Keller KL, Rolls BJ. Portion size can be used strategically to increase intake of vegetables and fruits in young children over multiple days: a cluster-randomized crossover trial. Am J Clin Nutr. 2022 Jan 11;115(1):272-283. doi: 10.1093/ajcn/nqab321. PMID 34550306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from three childcare centers in central Pennsylvania between November 2017 and March 2019
Groups:
- Con First, Then Add, Then Sub: Participants in the classrooms that received the three food proportionality interventions across the three periods in the order of Control, then Addition, then Substitution.
- Add First, Then Sub, Then Con: Participants in the classrooms that received the three food proportionality interventions across the three periods in the order of Addition, then Substitution, then Control.
- Sub First, Then Con, Then Add: Participants in the classroom that received the three food proportionality interventions across the three periods in the order of Substitution, then Control, then Addition.
- Con First, Then Sub, Then Add: Participants in the classroom that received the three food proportionality interventions across the three periods in the order of Control, then Substitution, then Addition.
- Add First, Then Con, Then Sub: Participants in the classroom that received the three food proportionality interventions across the three periods in the order of Addition, then Control, then Substitution.
- Sub First, Then Add, Then Con: Participants in the classroom that received the three food proportionality interventions across the three periods in the order of Substitution, then Addition, then Control.
Period: Study Week 1
Arm/Group | Con First, Then Add, Then Sub | Add First, Then Sub, Then Con | Sub First, Then Con, Then Add | Con First, Then Sub, Then Add | Add First, Then Con, Then Sub | Sub First, Then Add, Then Con
Started | 13 | 16 | 4 | 4 | 15 | 5
Completed | 13 | 15 | 4 | 4 | 12 | 5
Not Completed | 0 | 1 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 3 | 0
Period: Study Week 2
Arm/Group | Con First, Then Add, Then Sub | Add First, Then Sub, Then Con | Sub First, Then Con, Then Add | Con First, Then Sub, Then Add | Add First, Then Con, Then Sub | Sub First, Then Add, Then Con
Started | 13 | 15 | 4 | 4 | 12 | 5
Completed | 13 | 15 | 4 | 4 | 12 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Study Week 3
Arm/Group | Con First, Then Add, Then Sub | Add First, Then Sub, Then Con | Sub First, Then Con, Then Add | Con First, Then Sub, Then Add | Add First, Then Con, Then Sub | Sub First, Then Add, Then Con
Started | 13 | 15 | 4 | 4 | 12 | 5
Completed | 13 | 15 | 4 | 4 | 12 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Enrolled participants who completed the study
Arm/Group | Entire Study Population
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.4 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 6
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Differences in Food and Beverage Intake by Energy
Description: Differences in daily energy consumed of food and beverages, in kilocalories
Time Frame: Day 1-5 in weeks 1, 2, and 3
Measure: Mean (Standard Error); unit: kilocalories per day
Arm/Group | Control | Addition | Substitution
Number analyzed (Participants) | 53 | 53 | 53
kilocalories per day | 1059 (33) | 1118 (35) | 977 (34)
Statistical Analysis 1: Comparison: Control vs Addition vs Substitution; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Primary Outcome: Differences in Food and Beverage Intake by Weight
Description: Differences in daily weight consumed of food and beverages, in grams
Time Frame: Day 1-5 in weeks 1, 2, and 3
Measure: Mean (Standard Error); unit: grams per day
Arm/Group | Control | Addition | Substitution
Number analyzed (Participants) | 53 | 53 | 53
grams per day | 868 (35) | 955 (36) | 908 (35)
Statistical Analysis 1: Comparison: Control vs Addition vs Substitution; Test type: Superiority; p = 0.0015, Mixed Models Analysis

3. Primary Outcome: Differences in Food and Beverage Intake by Weight
Description: Differences in daily weight consumed of vegetables and fruit, in grams
Time Frame: Day 1-5 in weeks 1, 2, and 3
Measure: Mean (Standard Error); unit: grams per day
Arm/Group | Control | Addition | Substitution
Number analyzed (Participants) | 53 | 53 | 53
grams per day | 225 (15) | 296 (15) | 315 (15)
Statistical Analysis 1: Comparison: Control vs Addition vs Substitution; Test type: Superiority; p < 0.0001, Mixed Models Analysis

4. Secondary Outcome: Differences in Food and Beverage Intake by Energy Density
Description: Differences in daily energy density consumed of food and beverages, in kilocalories/gram
Time Frame: Day 1-5 in weeks 1, 2, and 3
Measure: Mean (Standard Error); unit: kilocalories/gram per day
Arm/Group | Control | Addition | Substitution
Number analyzed (Participants) | 53 | 53 | 53
kilocalories/gram per day | 1.29 (0.038) | 1.21 (0.039) | 1.14 (0.038)
Statistical Analysis 1: Comparison: Control vs Addition vs Substitution; Test type: Superiority; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Control: All participants during the Control condition
- Addition: All participants during the Addition condition
- Substitution: All participants during the Substitution condition
Arm/Group | Control | Addition | Substitution
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT03242863/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT03242863/Prot_SAP_002.pdf